## **Integrated Analysis Plan**

**Clinical Trial Protocol** 

Identification No.

MS201923-0007

Title

A Rollover Study to Provide Continued Treatment with M6620

Trial Phase

**Investigational Medicinal** 

Product(s)

M6620

Ι

Clinical Trial Protocol

Version

08 September 2017 / Version 2.0

**Integrated Analysis Plan** 

Author

**Coordinating Author** 

PPD , Merck PPD

Function Author(s) / Data Analyst(s)

PPD PPD

**Integrated Analysis Plan** 

**Date and Version** 

28 January 2019 / Version 1

**Integrated Analysis Plan** 

Reviewers

Function
PPD
PPD, Merck
PPD, Merck

Name PPD PPD PPD

#### Confidential

This document is the property of Merck KGaA, Darmstadt, Germany, or one of its affiliated companies. It is intended for restricted use only and may not - in full or part - be passed on, reproduced, published or used without express permission of Merck KGaA, Darmstadt, Germany or its affiliate.

Copyright © 2018 by Merck KGaA, Darmstadt, Germany or its affiliate. All rights reserved.

# **Approval Page**

**Integrated Analysis Plan:** MS201923-0007

A Rollover Study to Provide Continued Treatment with M6620

| Merck responsible | Date | Signature |
|-------------------|------------|---------------------|
| PPD | Via ELDORA | DO approval process |

## ATRi Transition Rollover Study

| 1 | Table of Contents | |
|---|---|---|
| Integrated Analy | sis Plan | 1 |
| Approval Page | 2 | |
| 1 | Table of Contents | 3 |
| 2 | List of Abbreviations and Definition of Terms | 4 |
| 3 | Modification History | 5 |
| 4 | Purpose of the Integrated Analysis Plan | 5 |
| 5 | Objectives and Endpoints | 5 |
| 6 | Overview of Planned Analyses | 5 |
| 7 | Changes to the Planned Analyses in the Clinical Trial Protocol | 5 |
| 8 | Protocol Deviations and Analysis Sets | 5 |
| 9 | General Specifications for Data Analyses | 6 |
| 10 | Trial Subjects | 6 |
| 10.1 | Disposition of Subjects and Discontinuations | 6 |
| 10.2 | Protocol Deviations | 6 |
| 11 | Demographics and Other Baseline Characteristics | 6 |
| 12 | Concomitant Medications/Procedures | 6 |
| 13 | Treatment Compliance and Exposure | 6 |
| 14 | Efficacy Analyses | 6 |
| 15 | Safety Analyses | 6 |
| 15.1 | Adverse Events | 7 |
| 15.2 | Clinical Laboratory Evaluation. | 7 |
| 15.3 | Vital Signs | 7 |
| 16 | References. | 7 |
| 17 | Appendices | 7 |

#### **ATRi Transition Rollover Study**

#### 2 List of Abbreviations and Definition of Terms

AE Adverse Event

eCRF Electronic Case Report Form

ENR Enrolled Analysis Set
IAP Integrated Analysis Plan

ICH International Conference on Harmonization

MedDRA Medical Dictionary for Regulatory Activities

NCI-CTCAE National Cancer Institute – Common Terminology Criteria for Adverse

**Events** 

SAE Serious Adverse Event SAF Safety Analysis Set

SDTM Study Data Tabulation Model

WHO-DD World Health Organization-Drug Dictionary

## **Modification History**

| Unique<br>Identifier for<br>Version | Date of IAP Version | Author | Changes from the Previous Version |
|---|---|---|---|
| 1.0 | 28Jan2019 | PPD | Initial version. |

## 4 Purpose of the Integrated Analysis Plan

The purpose of this Integrated Analysis Plan (IAP) is to document technical and detailed specifications for the presentation of data collected for protocol MS201923-0007.

The IAP is based upon Section 8 (Statistics) of the trial protocol and protocol amendments and is prepared in compliance with International Conference on Harmonization (ICH) E9.

### 5 Objectives and Endpoints

| | Objective | Endpoint | IAP section |
|---|---|---|---|
| Primary<br>Objective | To monitory safety of subjects that are on long-term treatment with M6620. | Occurrence adverse events (AEs) in subjects receiving M6620, graded according to National Cancer Institute Common Terminology Criteria for AEs (NCI-CTCAE) (Version 4.03), 28 days after the last administration of M6620. | 15.1 |

## **6** Overview of Planned Analyses

There are no interim analyses planned for this study. All final, planned analyses identified in the Clinical Trial Protocol and in this IAP will be performed only after the last subject has completed the study with all trial data in-house, all data queries resolved, and the database locked.

A data review meeting will be held prior to database lock. In addition, no database can be locked until this IAP has been approved.

# 7 Changes to the Planned Analyses in the Clinical Trial Protocol

Due to the small number of subjects on the study, no statistical analysis will be conducted, and the data will be presented in listings only.

## **8** Protocol Deviations and Analysis Sets

The following populations are defined per protocol.

Enrolled analysis set (ENR): All subjects who sign informed consent for this study.

**Safety analysis set (SAF):** All subjects who receive at least 1 dose of study drug in this study. Subjects will be analyzed according to the actual treatment they receive.

## 9 General Specifications for Data Analyses

All data will be listed as collected, and no derived datasets will be produced. All listings will be based upon the Study Data Tabulation Model (SDTM) datasets. Subjects will be listed according to the cohort in which they were continued from the previous study.

## Trial Subjects

### 10.1 Disposition of Subjects and Discontinuations

Subject disposition and treatment/trial discontinuation data will be listed as collected on the electronic case report form (eCRF).

#### 10.2 Protocol Deviations

All important deviations from inclusion/exclusion criteria will be listed.

### 11 Demographics and Other Baseline Characteristics

All demographic and baseline characteristics data will be listed as collected on the eCRF.

#### 12 Concomitant Medications/Procedures

Concomitant medications, as reported on the eCRF, will be listed according to the Anatomical Therapeutic Class (ATC) Level 2 text and preferred term as given from the current version of the World Health Organization-Drug Dictionary (WHO-DD) dictionary at time of database lock and noted as to whether they were ongoing at the time of study transition.

Concomitant procedures will be listed according to the reported name and standardized name as given from the current version of the Medical Dictionary for Regulatory Activities (MedDRA) dictionary at the time of database lock.

## 13 Treatment Compliance and Exposure

All exposure data will be listed, as collected on the eCRF, by the drug administered.

### 14 Efficacy Analyses

Not applicable.

#### 15 Safety Analyses

All safety data will be listed as collected on the eCRF.

#### **15.1** Adverse Events

All adverse events (AEs) will be listed according to the preferred term as given from the current version of the MedDRA dictionary at the time of database lock. All serious adverse events (SAEs) will be noted in the main AE listing, and a separate SAE listing will be produced.

# 15.2 Clinical Laboratory Evaluation

Clinical laboratory results will be listed with the applicable normal ranges along with flags for above/below normal range.

## 15.3 Vital Signs

All vitals sign results and subject weights will be listed as collected on the eCRF.

#### 16 References

Not applicable.

## 17 Appendices

Not applicable.